CLINICAL TRIAL: NCT00472459
Title: A Multicenter, Randomized Study of Photodynamic Therapy (PDT) With Metvix® 160 mg/g Cream in Immuno-compromised Patients With Non-melanoma Skin Cancer
Brief Title: Photodynamic Therapy (PDT) With Metvix® 160 Milligrams/Gram Cream in Organ Transplant Participants With Non-melanoma Skin Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PC T313/03
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-03

CONDITIONS: Actinic Keratosis; Warts; Basal Cell Carcinoma; Bowens Disease; Squamous Cell Carcinoma
Keywords: Non-melanoma skin cancer; Organ transplant recipients; Photodynamic therapy; Actinic keratosis
MeSH Terms: conditions — Keratosis, Actinic; Warts; Carcinoma, Basal Cell; Bowen's Disease; Carcinoma, Squamous Cell | interventions — Photochemotherapy; methyl 5-aminolevulinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metvix®-PDT (Treatment Area +Contralateral Control Area) (Experimental): Two contralateral areas (symmetrically) were identified with an area of 5*10-centimeter square, that is (i.e.), treatment and control area. Treatment area was treated with Metvix®-photodynamic therapy (PDT) 160 milligrams/gram (mg/g) cream, given as fractioned regimen consisting of two treatments one week apart on Weeks 0 and Week 1, additional single treatments were given at Months 3, 9, 15, 21 and 27. The contralateral control area was treated using lesion-specific treatment in accordance with the Investigator's preference (example, cryotherapy) at months 3, 9, 15, 21 and 27.
  Interventions: Procedure: Photodynamic therapy with Metvix 160 mg/g cream

INTERVENTIONS:
Procedure: Photodynamic therapy with Metvix 160 mg/g cream

SUMMARY:
Participants on immunosuppressive therapy, e.g., organ recipients, had higher occurrence of AK (Actinic Keratosis) than the untreated population. Keratotic lesions (i.e., AK lesions and warts) in this population were highly associated with development of SCC (Squamous Cell Carcinoma) also with 10 times higher mortality rate because of SCC than expected. The risk of developing skin cancer, predominantly SCC and BCC (Basal Cell Carcinoma), increased with graft survival time and the length of immunosuppressive treatment period.

The higher risk of developing skin malignancy and more aggressive skin malignancies in this population, indicated the need for early removal of these pre-malignant lesions.

In this study, two contralateral areas (5x10 cm^2) with skin lesions within the participant were compared. One area was received Metvix PDT at defined intervals and the other was received lesion specific treatment at the discretion of the investigator. The primary endpoint was the accumulated number of new lesions during the study and number of AK lesions that showed complete response 3 months after baseline. Secondary endpoints were number of BCC lesions that showed complete response, number of recurrent lesions, assessment of cosmetic outcome and safety.

DETAILED DESCRIPTION:
The treatment area (5x10 cm^2) was treated at baseline and at 3 ,9 and 15 months visits. At baseline, the area was treated with fractionated Metvix® PDT treatment consisting of two treatment one week apart and at 3 ,9 and 15 months visits with single Metvix® PDT treatment. The participants were evaluated for occurrence of new lesions, lesion response and recurrence at 3 (not recurrence),9,15,21, and 27 months visits. New and recurrent lesions in the treated area were treated with Metvix® PDT treatment. Lesions with partial response in the treated area were re-treated with Metvix® PDT and lesions with no response were treated with lesion specific treatment at the discretion of the investigator.

In the contralateral control area (5x10 cm^2), new and recurrent lesions and lesions in non-complete response were treated with lesion specific treatment at the discretion of the investigator at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Transplant recipients with at least 2 clinically diagnosed AK lesion and maximum 10 skin lesions (AK, BCC, SCC in situ and/or warts) in each of the two contralateral areas (diameter 5x10^2 cm) in the face, the scalp, the extremities or on the trunk/neck.
* Transplant recipients who previously were treated more than once for their skin lesions.
* Transplant recipients who had received immunosuppressive therapy for more than 3 years.
* Males or females above 18 years of age.
* Written informed consent.

Exclusion Criteria:

* Participants with more than 10 skin lesions (AK, BCC, SCC in situ, warts) in one of the two areas.
* Participants with SCC (not SCC in situ) in one of the two areas.
* Participants not previously treated or treated only once for their skin lesions.
* Participants with rosacea in one of the two areas.
* Participants with morphea form/highly infiltrating BCC
* Known allergy to methyl-amino levulinate, a similar compound or excipients of the cream
* Participation in other clinical studies either concurrently or within the last 30 days.
* Pregnant or breast-feeding (all women of child-bearing potential documented a negative pregnancy test and used the pill or IUD during the treatments and for at least one month thereafter).
* Conditions associated with a risk of poor protocol compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2003-07-25 (Actual); Primary Completion 2004-09-23 (Actual); Study Completion 2006-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Marie Wennberg, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (11):
- Denmark (2):
  - Department of Dermatology, Århus Amysygehus, Aarhus
  - Department of Dermatology, Roskilde Amysygehus, Roskilde
- Germany (2):
  - Klinik für Dermatologie, Venerologie und Allergologie, Campus Charité Mitte, Berlin
  - Hautklinik Linden, Hanover
- Norway (2):
  - Department of Dermatology, Rikshospitalet, Oslo
  - Department of Dermatology, St. Olavs Hospital, Trondheim
- Sweden (3):
  - Department of Dermatology, Sahlgrenska University Hospital, Gothenburg
  - Department of Dermatology, Karolinska University Hospital, Huddinge, Stockholm
  - Department of Dermatology, Uppsala University Hospital, Uppsala
- United Kingdom (2):
  - Dermatology Department, Manchester Royal Infirmary, Manchester
  - Portsmouth Dermatology Centre, St Mary's Hospital, Portsmouth

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 countries (Denmark, Germany, Norway, Sweden, and United Kingdom) between 25 July 2003 to 14 July 2006.
Pre-assignment Details: A total of 82 participants were randomized in the study, of which 81 participants were treated on one side of the participant (Treatment area) with Metvix®-PDT and other side of the participants (Contralateral Control Area).
Units Other Than Participants: Skin lesions
Groups:
- Metvix®- PDT (Treatment Area): Two contralateral areas (symmetrically) were identified with an area of 5*10-centimeter square, i.e., treatment and control area. Treatment area was treated with Metvix®-photodynamic therapy (PDT) 160 mg/g cream, given as fractioned regimen consisting of two treatments one week apart on Weeks 0 and Week 1, additional single treatments were given at Months 3, 9, 15, 21 and 27.
- Contralateral Control Area: The contralateral control area was treated using lesion-specific treatment in accordance with the investigator's preference (example, cryotherapy) at months 3, 9, 15, 21 and 27.
Period: Overall Study
Arm/Group | Metvix®- PDT (Treatment Area) | Contralateral Control Area
Started | 81; 485 Skin lesions | 81; 422 Skin lesions
Completed | 55; 476 Skin lesions | 55; 413 Skin lesions
Not Completed | 26; 9 Skin lesions | 26; 9 Skin lesions
Not completed — Adverse Event | 13 | 13
Not completed — Withdrawal by Subject | 5 | 5
Not completed — Protocol Violation | 3 | 3
Not completed — Heavy workload, Not satisfied, Squamous Cell Carcinoma | 4 | 4
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population included all treated participants. As per planned analysis unique participants baseline was not analysed, only overall participant data was analysed and reported.
Groups:
- All Study Participants: All participants were transplant recipients who had received immune suppressive therapy for at least 3 years and had skin lesions in each of two symmetrical contralateral areas on the face, scalp, extremities or trunk/neck received Metrvix®-PDT on one side of patient (treatment area) given as fractionated regimen on Week 0, Week 1, 3 months, 9 months and 15 months followed by other side of the patients selected area (Contralateral Control Area) was treated using lesion-specific treatment in accordance with the Investigator's preference.
Arm/Group | All Study Participants
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 81

OUTCOME MEASURES:

1. Primary Outcome: Number of Accumulated New Skin Lesions at Month 3
Description: A new lesion was defined as a visible new lesion of any size after the Baseline. New skin lesions accumulated were sum of actinic keratoses (AK) lesions, basal cell carcinoma (BCC) lesions, squamous cell carcinoma (SCC) lesions and warts in treated area and contralateral control area (symmetrically). Number of accumulated new skin lesions at Month 3 were reported.
Time Frame: At Month 3
Population: Intent-to-Treat (ITT) Population included all treated participants. Here, 'Overall Number of Units Analyzed' reflects the total number of skin lesions analyzed in each Arm.
Measure: Number; unit: new skin lesions
Units Other Than Participants: skin lesions
Arm/Group | Metvix®- PDT (Treatment Area) | Contralateral Control Area
Number analyzed (Participants) | 81 | 81
Number analyzed (skin lesions) | 476 | 413
new skin lesions | 65 | 103
Statistical Analysis 1: Comparison: Metvix®- PDT (Treatment Area) vs Contralateral Control Area; Test type: Non-Inferiority — Participant's number of new skin lesions between treated and contralateral control area were evaluated using a paired t-test for lesions of any type as well as stratified by lesion type; p = 0.0120, t-test, 2 sided; Mean Difference (Final Values) = 0.514, 95% CI 2-sided [0.116 to 0.911] — The 95 % confidence intervals for the lesion complete response rates and lesion recurrence rates were estimated using the method of Clopper and Pearson

2. Primary Outcome: Number of Accumulated New Skin Lesions at Month 9
Description: A new lesion was defined as a visible new lesion of any size after the Baseline. New skin lesions accumulated were sum of AK lesions, BCC lesions, SCC lesions and warts in treated area and contralateral control area (symmetrically). Number of accumulated new skin lesions at Month 9 were reported.
Time Frame: At Month 9
Population: ITT Population included all treated participants. Here, 'Overall Number of Units Analyzed' reflects the total number of skin lesions analyzed in each Arm.
Measure: Number; unit: new skin lesions
Units Other Than Participants: skin lesions
Groups:
- Metvix®-PDT (Treatment Area): Two contralateral areas (symmetrically) were identified with an area of 5*10-centimeter square, i.e., treatment and control area. Treatment area was treated with Metvix®-photodynamic therapy (PDT) 160 mg/g cream, given as fractioned regimen consisting of two treatments one week apart on Weeks 0 and Week 1, additional single treatments were given at Months 3 ,9, 15, 21 and 27.
Arm/Group | Metvix®-PDT (Treatment Area) | Contralateral Control Area
Number analyzed (Participants) | 81 | 81
Number analyzed (skin lesions) | 476 | 413
new skin lesions | 92 | 85
Statistical Analysis 1: Comparison: Metvix®-PDT (Treatment Area) vs Contralateral Control Area; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.1761, t-test, 2 sided; Mean Difference (Final Values) = 0.413, 95% CI 2-sided [-0.190 to 1.016]

3. Primary Outcome: Number of Accumulated New Skin Lesions at Month 15
Description: A new lesion was defined as a visible new lesion of any size after the Baseline. New skin lesions accumulated were sum of AK lesions, BCC lesions, SCC lesions and warts in treated area and contralateral control area (symmetrically). Number of accumulated new skin lesions at Month 15 were reported.
Time Frame: At Month 15
Population: as for outcome 2
Measure: Number; unit: new skin lesions
Units Other Than Participants: skin lesions
Groups:
- Metvix®-PDT (Treatment Area): Two contralateral areas (symmetrically) were identified with an area of 5*10-centimeter square, i.e., treatment and control area. Treatment area was treated with Metvix®-photodynamic therapy (PDT) 160 mg/g cream, given as fractioned regimen consisting of two treatments one week apart on Weeks 0 and Week 1, additional single treatments were given at Months 3, 9, 15, 21 and 27.
- Contralateral Control Area: The contralateral control area was treated using lesion-specific treatment in accordance with the investigator's preference (e.g., cryotherapy) at months 3, 9, 15, 21 and 27.
Arm/Group | Metvix®-PDT (Treatment Area) | Contralateral Control Area
Number analyzed (Participants) | 81 | 81
Number analyzed (skin lesions) | 476 | 413
new skin lesions | 73 | 87
Statistical Analysis 1: Comparison: Metvix®-PDT (Treatment Area) vs Contralateral Control Area; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.1183, t-test, 2 sided; Mean Difference (Final Values) = 0.600, 95% CI 2-sided [-0.156 to 1.357]

4. Primary Outcome: Number of Accumulated New Skin Lesions at Month 21
Description: A new lesion was defined as a visible new lesion of any size after the Baseline. New skin lesions accumulated were sum of AK lesions, BCC lesions, SCC lesions and warts in treated area and contralateral control area (symmetrically). Number of accumulated new skin lesions at Month 21 were reported.
Time Frame: At Month 21
Population: as for outcome 2
Measure: Number; unit: new skin lesions
Units Other Than Participants: skin lesions
Arm/Group | Metvix®-PDT (Treatment Area) | Contralateral Control Area
Number analyzed (Participants) | 81 | 81
Number analyzed (skin lesions) | 476 | 413
new skin lesions | 55 | 47
Statistical Analysis 1: Comparison: Metvix®-PDT (Treatment Area) vs Contralateral Control Area; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.2322, t-test, 2 sided; Mean Difference (Final Values) = 0.493, 95% CI 2-sided [-0.323 to 1.309]

5. Primary Outcome: Number of Accumulated New Skin Lesions at Month 27
Description: A new lesion was defined as a visible new lesion of any size after the Baseline. New skin lesions accumulated were sum of AK lesions, BCC lesions, SCC lesions and warts in treated area and contralateral control area (symmetrically). Number of accumulated new skin lesions at Month 27 were reported.
Time Frame: At Month 27
Population: as for outcome 2
Measure: Number; unit: new skin lesions
Units Other Than Participants: skin lesions
Arm/Group | Metvix®- PDT (Treatment Area) | Contralateral Control Area
Number analyzed (Participants) | 81 | 81
Number analyzed (skin lesions) | 476 | 413
new skin lesions | 38 | 52
Statistical Analysis 1: Comparison: Metvix®- PDT (Treatment Area) vs Contralateral Control Area; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.1286, t-test, 2 sided; Mean Difference (Final Values) = 0.680, 95% CI 2-sided [-0.202 to 1.562]

6. Primary Outcome: Number of AK Lesions That Showed Complete Response at Month 3
Description: Complete response was defined as the complete disappearance of the lesion. The AK lesions were graded as grade 1(mild); slightly palpable AK, better felt than seen, grade 2 (moderate); moderately thick AK, easily felt and seen, and grade 3 (severe); very thick and/or obvious AK. Mantel-Haenszel weighted difference was used to calculate number of AK lesions that showed complete response.
Time Frame: At Month 3
Population: ITT Population included all treated participants. Here, 'Overall Number of Units Analyzed' reflects the total number of AK lesions analyzed in each Arm.
Measure: Number; unit: skin lesions
Units Other Than Participants: skin lesions
Arm/Group | Metvix®-PDT (Treatment Area) | Contralateral Control Area
Number analyzed (Participants) | 81 | 81
Number analyzed (skin lesions) | 427 | 361
skin lesions | 296 | 240

7. Primary Outcome: Number of AK Lesions That Showed Complete Response at Month 9
Description: as for outcome 6
Time Frame: At Month 9
Population: as for outcome 6
Measure: Number; unit: skin lesions
Units Other Than Participants: skin lesions
Arm/Group | Metvix®-PDT (Treatment Area) | Contralateral Control Area
Number analyzed (Participants) | 81 | 81
Number analyzed (skin lesions) | 427 | 361
skin lesions | 311 | 262

8. Primary Outcome: Number of AK Lesions That Showed Complete Response at Month 15
Description: as for outcome 6
Time Frame: At Month 15
Population: as for outcome 6
Measure: Number; unit: skin lesions
Units Other Than Participants: skin lesions
Arm/Group | Metvix®-PDT (Treatment Area) | Contralateral Control Area
Number analyzed (Participants) | 81 | 81
Number analyzed (skin lesions) | 427 | 361
skin lesions | 286 | 236

9. Primary Outcome: Number of AK Lesions That Showed Complete Response at Month 21
Description: as for outcome 6
Time Frame: At Month 21
Population: as for outcome 6
Measure: Number; unit: skin lesions
Units Other Than Participants: skin lesions
Arm/Group | Metvix®-PDT (Treatment Area) | Contralateral Control Area
Number analyzed (Participants) | 81 | 81
Number analyzed (skin lesions) | 427 | 361
skin lesions | 275 | 224

10. Primary Outcome: Number of AK Lesions That Showed Complete Response at Month 27
Description: as for outcome 6
Time Frame: At Month 27
Population: as for outcome 6
Measure: Number; unit: skin lesions
Units Other Than Participants: skin lesions
Arm/Group | Metvix®-PDT (Treatment Area) | Contralateral Control Area
Number analyzed (Participants) | 81 | 81
Number analyzed (skin lesions) | 427 | 361
skin lesions | 265 | 206

11. Secondary Outcome: Number of BCC Lesions That Showed Complete Response
Description: Complete response was defined as the complete disappearance of the lesion. BCC lesions were characterized as superficial: ill-defined red scaly macule; could increase in size to form crusted, occasionally ulcerated, scaly erythematous patches, but never indurated and nodular: flesh-colored, cream to pink, waxy papule with prominent surface telangiectasias; as the lesions grow, central erosion or ulceration and crusting occur, surrounded by a pearly, rolled, translucent border. Number of BCC lesions that showed complete response was reported.
Time Frame: At Months 3, 9, 15, 21 and 27
Population: ITT Population included all treated participants. Here, 'Overall Number of Units Analyzed' reflects the total number of BCC lesions analyzed in each Arm.
Measure: Number; unit: skin lesions
Units Other Than Participants: skin lesions
Arm/Group | Metvix®-PDT (Treatment Area) | Contralateral Control Area
Number analyzed (Participants) | 81 | 81
Number analyzed (skin lesions) | 2 | 2
skin lesions
  Month 3 | 1 | 2
  Month 9 | 0 | 2
  Month 15 | 0 | 2
  Month 21 | 0 | 2
  Month 27 | 1 | 2

12. Secondary Outcome: Number of Recurrent Lesions
Description: Recurrence of lesions was defined as reappearance of previously treated and eradicated lesions and was verified by histology in accordance with local hospital practice.
Time Frame: At Months 9, 15, 21 and 27
Population: ITT population included all participants who were enrolled and treated at baseline. Here, 'Overall Number of Units Analyzed' reflects the total number of skin lesions analyzed in each Arm.
Measure: Number; unit: skin lesions
Units Other Than Participants: skin lesions
Groups:
- Metvix®-PDT: Two contralateral areas (symmetrically) were identified with an area of 5*10-centimeter square, i.e., treatment and control area. Treatment area was treated with Metvix®-photodynamic therapy (PDT) 160 mg/g cream, given as fractioned regimen consisting of two treatments one week apart on Weeks 0 and Week 1, additional single treatments were given at Months 3, 9, 15, 21 and 27.
- Placebo-PDT: The contralateral control area was treated using lesion-specific treatment in accordance with the investigator's preference (example, cryotherapy) at months 3, 9, 15, 21 and 27.
Arm/Group | Metvix®-PDT | Placebo-PDT
Number analyzed (Participants) | 81 | 81
Number analyzed (skin lesions) | 476 | 413
skin lesions
  Month 9: number analyzed (skin lesions) | 321 | 272
  Month 9 | 24 | 14
  Month 15: number analyzed (skin lesions) | 341 | 303
  Month 15 | 31 | 20
  Month 21: number analyzed (skin lesions) | 310 | 276
  Month 21 | 12 | 8
  Month 27: number analyzed (skin lesions) | 303 | 260
  Month 27 | 10 | 4

13. Secondary Outcome: Number of Participants With Overall Cosmetic Outcome Assessed by Investigator and Participants
Description: Overall cosmetic outcome for the two contralateral areas (treatment and contralateral control) with an area of 5 by 10 cm^2 was assessed with regards to either absence or presence of all signs or symptoms or the presence of at least one of the signs or symptoms; scarring, atrophy, depigmentation, redness and fibrosis by both investigator and participant. Parameters were assessed for each area were hypopigmentation, hyperpigmentation, scar formation and tissue defect. The occurrence of these parameters was graded as none, slight, or obvious. Cosmetic outcome was presented as number of participants in each category (none, slight, obvious) for each variable assessed (hypopigmentation, hyperpigmentation, scar formation, tissue defect).
Time Frame: At Month 27
Population: ITT-population. Here, "overall number of participants analyzed" signifies number of participants evaluable for this outcome measure and "number analyzed" signifies participants evaluable for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Metvix®-PDT (Treatment Area) | Contralateral Control Area
Number analyzed (Participants) | 55 | 55
Participants
  Hyperpigmentation (Assessor- Investigator): None | 50 | 50
  Hyperpigmentation (Assessor- Investigator): Slight/Obvious | 5 | 5
  Hyperpigmentation (Assessor- Participant): None: number analyzed (Participants) | 54 | 54
  Hyperpigmentation (Assessor- Participant): None | 51 | 52
  Hyperpigmentation (Assessor- Participant): Slight/Obvious | 3 | 2
  Hypopigmentation (Assessor- Investigator): None | 46 | 27
  Hypopigmentation (Assessor- Investigator): Slight/Obvious | 9 | 28
  Hypopigmentation (Assessor- Participant): None: number analyzed (Participants) | 54 | 54
  Hypopigmentation (Assessor- Participant): None | 49 | 36
  Hypopigmentation (Assessor- Participant): Slight/Obvious | 5 | 18
  Scar formation (Assessor- Investigator): None | 48 | 42
  Scar formation (Assessor- Investigator): Slight/Obvious | 7 | 13
  Scar formation (Assessor- Participant: None: number analyzed (Participants) | 54 | 54
  Scar formation (Assessor- Participant: None | 47 | 40
  Scar formation (Assessor- Participant): Slight/Obvious | 7 | 14
  Tissue defect (Assessor- Investigator): None | 52 | 53
  Tissue defect (Assessor- Investigator): Slight/Obvious | 3 | 2
  Tissue defect (Assessor- Participant): None: number analyzed (Participants) | 54 | 54
  Tissue defect (Assessor- Participant): None | 51 | 53
  Tissue defect (Assessor- Participant): Slight/Obvious: number analyzed (Participants) | 54 | 54
  Tissue defect (Assessor- Participant): Slight/Obvious | 3 | 1

14. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: From Baseline up to Month 27
Population: Safety Population that included in the study and received Metvix® cream were included in safety evaluation.
Measure: Count of Participants; unit: Participants
Groups:
- Metvix®-PDT: Two contralateral areas (symmetrically)were identified with an area of 5*10-centimeter square,i.e., treatment and control area. Treatment area was treated with Metvix® PDT 160mg/g cream, given as fractioned regimen consisting of two treatments one week apart on Weeks 0 and Week 1, additional single treatments given were given at Months 3, 9, 15, 21 and 27. Adverse Events localized to the treatment area are reported.
- Contralateral Control Area: The contralateral control area was treated using lesion-specific treatment in accordance with the investigator's preference (example, cryotherapy) at months 3, 9, 15, 21and 27. Adverse Events localized to the contralateral Control Area.
- Not Applicable: Participants none of the area were assigned to either of treatment. All Adverse Events, including those that affected participants as a whole (systemic events).
Arm/Group | Metvix®-PDT | Contralateral Control Area | Not Applicable
Number analyzed (Participants) | 81 | 81 | 81
Participants
  Participants with AE | 61 | 39 | 27
  Participants with SAE | 4 | 1 | 26

ADVERSE EVENTS:
Time Frame: Adverse events data were reported from the first treatment up to the 27-month follow up period.
Description: Safety population that included in the study and received Metvix® cream were included in safety evaluation. Data on all serious and non-serious Adverse Events experienced by participants were collected, irrespective of the event's relation to the treatment area. Participants with systemic Adverse Events were not considered at risk for these events in the Treatment area and contralateral control area arms since those arms were limited to the analysis of localized events.
Groups:
- All Study Participants: Participants none of the area were assigned to either of treatment. All Adverse Events, including those that affected participants as a whole (systemic events).
Arm/Group | Metvix®-PDT | Contralateral Control Area | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/81 | 6/81
Serious Adverse Events (participants affected / at risk) | 4/81 | 1/81 | 26/81
Other Adverse Events (participants affected / at risk) | 61/81 | 39/81 | 27/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metvix®-PDT (N=81) | Contralateral Control Area (N=81) | All Study Participants (N=81)
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 1 (2) | 3 (4)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Thyroid Gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Urosepsis (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Parathyroidectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Renal Transplant (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Wound Secretion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Knee Arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Calcus Urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Postoperative Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Post Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Neoplasm Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal Impairement (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fluid Overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Complications of Transplanted Kidney (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Herpes Simplex Ophthalmic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metvix®-PDT (N=81) | Contralateral Control Area (N=81) | All Study Participants (N=81)
Erythema (Skin and subcutaneous tissue disorders) | 53 | 22 | 0
Pain of Skin (Skin and subcutaneous tissue disorders) | 44 | 32 | 1
Scab (Skin and subcutaneous tissue disorders) | 19 | 14 | 0
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 8 | 1 | 0
Skin Oedema (Skin and subcutaneous tissue disorders) | 7 | 3 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 2 | 10 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 22
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 5
Angioneurotic Oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Leukocytoclastic Vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin Nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Stasis Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other